CLINICAL TRIAL: NCT00912470
Title: Genetic Vascular Risk Factors and Ocular Blood Flow in Patients With Progressive Open Angle Glaucoma (OAG)-a Longitudinal Prospective Study
Brief Title: Progressive Open Angle Glaucoma (OAG) and Ocular Blood Flow
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Deparment of clinical pharmacology, Medical university of Vienna
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPHT-020706
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2014-11-21 (Estimated); Status verified 2014-11

CONDITIONS: Open Angle Glaucoma
Keywords: genetic vascular risc factors; ocular blood flow; progressive glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: ocular blood flow measurement — Retinal blood flow (with scanning laser Doppler flowmetry, laser Doppler velocimetry + retinal vessel analyzer) each measurement once on the study eye
  Choroidal blood flow (with laser Doppler flowmetry, laser interferometry, pneumotonometry)
  Frequency distribution of alleles of genetic markers for NOS3, more precisely eNOS -786CC polymorphism and of ET-1 (EDN1), and the receptors ETA (EDNRA), more precisely EDN1/+138/ex1 del/ins, EDN1/K198N, EDNRA/C+1222T, EDNRA/C+70G polymorphisms
  Other Names: Blood sample for Frequency distribution of alleles

SUMMARY:
The purpose of this study is to assess the correlation of vascular parameters, including genetic factors as well as ocular blood flow parameters against the progression rate of glaucomatous damage in patients with progressive OAG.

DETAILED DESCRIPTION:
Glaucoma is one of the most common causes of blindness in the industrialized nations. For a long time glaucoma has been defined as a disease in which high intraocular pressure (IOP) leads to irreversible optic disc damage and subsequent visual field loss. However, recent investigations show that IOP is not the only factor that is involved in the glaucomatous process leading to retinal ganglion cell death. The role of vascular factors in the pathogenesis of glaucoma has recently received much attention based on animal experiments and epidemiological studies. Genes with products that are involved in the regulation of blood flow to ocular tissues may also be considered plausible candidates as a contributory factor in the development of glaucoma. Little is, however, known about a potential association between glaucomatous optic neuropathy and glaucomatous visual field defects and optic nerve head blood flow in patients with progressive open angle glaucoma (OAG). The current study seeks to gain insight into this association by assessing ocular blood flow parameters with a number of noninvasive technologies.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 40 years
* Unilateral or bilateral primary open angle glaucoma (POAG) or normal tension glaucoma (NTG) with visual defect, marked by an AGIS score (1994; 1. Study design and methods and baseline characteristics of study patient) of at least 1 but not more than 16 at the screening visit
* At least 3 reliable visual field tests in the eye that will be studied
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Best-corrected visual acuity of 20/40 or better, spherical refraction within ± 3.0 diopters and cylinder correction within ± 3.0 diopters

Exclusion Criteria:

* Evidence of secondary glaucoma, pseudoexfoliation, pigmentary dispersion
* Any form of retinal or neuroophthalmological disease that could result in visual field defects.
* Mean IOP > 30 mmHg, or any IOP > 35 mmHg in at least one eye
* History of acute angle closure
* Closed or barely open anterior chamber angle
* Topical or systemical/oral therapy with steroids
* Standard deviation of visual field testing > 10
* Ocular inflammation or infection within the last three months
* Intraocular surgery or argon laser trabeculoplasty within the last six months
* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks
* Ametropia > 3 dpt

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-05; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Optic nerve head blood flow (scanning laser Doppler flowmetry, laser Doppler flowmetry). | up to 6 years.

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Garhöfer, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Vienna, Austria